CLINICAL TRIAL: NCT06674226
Title: Effects of Ciprofol on Postoperative Delirium and Outcomes in Elderly Patients Undergoing Major Thoracic Surgery: a Multicentre, Prospective, Single-blind, Randomized Controlled Study
Brief Title: Effects of Ciprofol on Postoperative Delirium and Outcomes in Elderly Patients Undergoing Major Thoracic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wang Tianlong (Other)
Collaborators: Xiangya Hospital of Central South University (Other); The Third Xiangya Hospital of Central South University (Other); The First Hospital of Hebei Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); Tongji Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor-Investigator, Wang Tianlong, professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Linyanshen[2024]201-002
Record Dates: First submitted 2024-10-31; First posted 2024-11-05 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Delirium (POD)
MeSH Terms: conditions — Emergence Delirium | interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ciprofol group (Experimental): Interventions:
  Drug:Ciprofol
  Interventions: Drug: Ciprofol
- Propofol group (Active Comparator): Drug:Propofol
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ciprofol — 0.25mg/kg for anesthesia induction ＋0.25~1.5 mg/kg/h for maintenance
  Arms: Ciprofol group
Drug: Propofol — 1.0mg/kg for induction ＋1 ~ 6mg/kg/h for maintenace
  Arms: Propofol group

SUMMARY:
There are many factors that make elderly patients prone to POD. On the basis of these factors, surgery and anesthesia can increase the incidence of POD in elderly patients. Deep depth of intraoperative anesthesia and persistent hypotension may increase the risk of POD occurrence in elderly patients. So far, no specific POD prevention method has been found. In recent years, a large number of studies on POD have brought forward more new views on its pathogenesis, prevention and treatment. There is insufficient evidence to recommend specific anesthetic agents and dosages to reduce the risk of POD in elderly patients, and only low-quality evidence to recommend propofol. At present, it is considered that the best way to reduce postoperative delirium is perioperative risk management, to evaluate high-risk patients or patients undergoing high-risk surgery as extensive as possible, and to quantify their risk of postoperative delirium. Effective measures include depth management of anesthesia, multi-modal analgesia management, and optimization of drug intervention.

Ciprofol is a class 1 innovative drug independently developed by China and with global independent intellectual property rights. Ciprofol has been widely used in anesthesiology and critical care medicine. The pre-market phase I-III and post-market data showed that during the induction and maintenance of general anesthesia, Ciprofol had less impact on hemodynamics and more stable anesthesia depth than propofol. Relevant studies have shown that Ciprofol can reduce the risk of hypotension, and can provide better brain oxygenation and more stable intraoperative hemodynamics than propofol. At present, the influence of different sedative drugs on POD incidence in elderly patients remains to be studied. Therefore, we will apply Ciprofol or propofol in elderly patients undergoing thoracic surgery to observe their influence on POD incidence and provide reference for clinical use.

DETAILED DESCRIPTION:
This study was a prospective, single-blinded, randomized controlled study. Elderly patients (≥65 years old) who were to receive elective thoracoscopic lobectomy and pulmonary segmentation under general anesthesia and whose estimated time of anesthesia (from the beginning of anesthesia to the end of surgery) was ≥2 hours were enrolled into this study, and were randomly divided according to 1:1, namely the ciprofol group and the propofol group. Study data of patients were recorded before surgery, during surgery, 7 days after surgery or before discharge.Primary end point: Incidence of postoperative delirium(Incidence of delirium on the first to seventh day after surgery or to the day of discharge (whichever occurs first)).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years old, gender unlimited;
* Selective thoracoscopic lobectomy and segmental lung resection were performed, and the estimated time of anesthesia (from the beginning of anesthesia to the end of surgery) was ≥2 hours;
* ASA score is Grade I ~III; (Annex 1)
* A BMI of 18.5 to 29.9 kg/m2 [BMI= weight (Kg)/height (m) 2] (2013 U.S. Guidelines for the Management of Overweight and Obesity in Adults);
* Postoperative hospital stay more than 72 hours;
* Ethical, patients voluntarily take the test and sign the informed consent.

Exclusion Criteria:

* Emergency surgery; Hypovolemia, shock or coma;
* In addition to general intravenous anesthesia, other anesthesia methods should be combined, such as inhalation anesthesia, epidural anesthesia, peripheral nerve block, etc., but it is not necessary to exclude patients with local infiltration of local anesthetic incision;
* Serious cardiovascular disease, including a history of myocardial infarction within 6 months, bradycardia (resting heart rate < 50 beats/min); Patients with hypertension whose blood pressure is not satisfactorily controlled (seated systolic blood pressure ≥160 mmHg during screening, and/or diastolic blood pressure ≥100 mmHg during screening); Sitting systolic blood pressure ≤90 mmHg during the screening period; A history of severe heart valve disease.
* Abnormal liver function, AST and/or ALT≥2.5×ULN, TBIL≥1.5×ULN;
* Abnormal renal function, urea or urea nitrogen ≥1.5×ULN, blood creatinine greater than the upper limit of normal;
* Glycated hemoglobin (HbA1c) ≥ 8.5%, fasting blood glucose ≥180 mg/dl (10 mmol/L), blood glucose ≥270mg/dl (15mmol/L) 1 hour after meals, or blood glucose ≥216 mg/dl (12mmol/L) 2 hours after meals;
* Patients with type I and type II expiratory failure
* Preoperative anemia (Hb≤90 g/L), thrombocytopenia (PLT≤80×109/L), hypoproteinemia (Alb≤30 g/L);
* A history of drug use and/or alcohol abuse within the 2 years prior to screening, with alcohol abuse being an average consumption of more than 2 units of alcohol per day (1 unit =360 mL beer or 150 mL of 45 mL liquor or wine with an alcohol concentration of 40%);
* Patients with neurological diseases (stroke, Alzheimer's disease, Parkinson's disease, mental illness, myasthenia grave, etc., within 6 months), psychiatric diseases (schizophrenia, mania, bipolar disorder, insanity, etc.), long-term history of taking psychiatric drugs and cognitive impairment (using the simple mental State Assessment Form (MMSE scale (Annex 2));
* Patients who take sedative sleeping drugs and antiepileptic drugs for a long time;
* Allergic to the investigational drug or contraindicated;
* Participated in other drug clinical trials as a subject within the last 3 months;
* Patients who refused or were unable to cooperate with the study;
* Other conditions that the investigator considers inappropriate to participate in this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | up to the seventh day after surgery or on the day of discharge (whichever occurs first).
  Incidence of delirium on the first to seventh day after surgery or on the day of discharge (whichever occurs first).

SECONDARY OUTCOMES:
Incidence of Emergence delirium | from the onset of extubation to departure of the PACU
  Delirium occurred from the onset of extubation to departure of the PACU was assessed using the CAM-ICU scale by a trained accessor who was not aware of this grouping
The incidence of combined adverse events during induction and maintenance of anesthesia; | During the intervention
Duration of intraoperative hypotension | During the intervention
  Hypotension is defined as invasive MAP<65mmHg or <80% of baseline value.
Minimum mean intraoperative arterial pressure | During the intervention
Duration of WLi < 40 | During the intervention
Other adverse events identified during the follow-up period, except POD | up to the seventh day after surgery or on the day of discharge (whichever occurs first).
Length of stay | Perioperatively
First exhaust time | up to the seventh day after surgery or on the day of discharge (whichever occurs first).
Postoperative first time to taking food | up to the seventh day after surgery or on the day of discharge (whichever occurs first).

CONTACTS AND LOCATIONS:
Overall Officials: Tianlong Wang, Doctor, Principal Investigator — Xuanwu Hospital, Beijing
Locations (8):
- China (8):
  - Xuanwu Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Jinan University, Guangzhou, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tongji Hospital, Wuhan, Hubei
  - The third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: After the article is published, contact the corresponding author to obtain

REFERENCES:
- [Derived] Hong P, Liu Q, Ouyang W, Luo A, Wang E, Gu X, Wang L, Chen S, Wang H, Xiao W, Wang T. Effects of ciprofol on postoperative delirium and outcomes in older patients undergoing major thoracic surgery: protocol for a multicentre, prospective, single-blinded, randomised controlled study. BMJ Open. 2025 Aug 19;15(8):e105818. doi: 10.1136/bmjopen-2025-105818. PMID 40829819